CLINICAL TRIAL: NCT03361462
Title: Community-based Mental Wellness Project for Adolescents and Adults: Joyful Adventure Day - A Pilot Project
Brief Title: Joyful Adventure Day for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Boys' and Girls' Clubs Association of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Daniel Sai-Yin Ho, Associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPH-MHP-BGCA01
Record Dates: First submitted 2017-11-27; First posted 2017-12-04 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Mental Health Wellness 1
Keywords: Sharing; Mind; Enjoyment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Two joyful adventure days in the form of physical activities and competitions with adventure games and short interactive talk on SME.
  Interventions: Behavioral: Joyful Adventure Day
- Waitlist control group (No Intervention): The intervention won't be provided during evaluation period and will be provided after the evaluation period

INTERVENTIONS:
Behavioral: Joyful Adventure Day — Participants will participate in two joyful adventure days with adventure games and a short talk on SME (Sharing, Mind, Enjoyment) focusing on positive thinking and understanding of adolescent mental health problem (in particular the anxiety disorders) and mental well-being; provide physical activity diary, such as "Zero-time Exercise" after 1st session of adventure day, and invite family members / peers to join the competition at the 2nd session.
  Arms: Intervention group

SUMMARY:
Joyful Adventure Day - A Pilot Project is part of the Community-based Mental Wellness Project for Adolescents and Adults, which aims at promoting Sharing, Mind and Enjoyment (SME) and enhancing mental wellbeing. The Mental Wellness Project is financially supported by the Health Care and Promotion Fund from Food and Health Bureau and led by the School of Public Health, University of Hong Kong (HKU). Joyful Adventure Day - A Pilot Project aims to promote the SME related behaviors of adolescents through intervention of physical activities, and to promote their happiness, well-being and mental health knowledge.

DETAILED DESCRIPTION:
A cluster randomized controlled trial design will be adopted. The Project will organize two joyful adventure days in secondary schools in the form of physical activities and competitions with the following activities:

* Fitness assessment (enjoyment) and in-door games, which will be designed, supervised and supported by experienced social workers;
* Short interactive talk on SME, positive thinking and understanding of adolescent mental health problem (in particular the anxiety disorders) and mental well-being;
* Issue achievement / improvement stickers to students, and attractive prizes to the 10 fittest students by chairperson / members of Parent-Teacher Association (sharing);
* Provide physical activity diary after 1st session of adventure day, and invite family members / peers to join the competition at the 2nd session.

The major subjects of Joyful Adventure Day Pilot Project RCT study are 200-300 students. 3 schools will be included in the evaluation. The classes in the same school will either be assigned into intervention group or waitlist control group (the intervention won't be provided during evaluation period and will be provided after the evaluation period.).

There will then be 4 assessments (pre-intervention, immediate post intervention, one month and three months after baseline) to evaluate the effects of the intervention programme. In the assessments, students will be asked to complete questionnaires to measure the changes in fitness enjoyment, physical activity frequency, happiness, well-being and knowledge and attitude towards mental health. The satisfaction towards the intervention, as well as the level of participation and ratings for the intervention will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Students (major subjects): (Intervention group and waitlist control group)

  1. Chinese speaking
  2. Intact verbal and hearing abilities for interpersonal communication
  3. Reading and writing abilities for questionnaire completion
  4. Secondary school students
* Parents: (Intervention group)

  1. Chinese speaking
  2. Intact verbal and hearing abilities for interpersonal communication
  3. Reading and writing abilities for questionnaire completion
  4. With at least one secondary school child
* School principals/teachers/community partners: (Intervention group)

  1. Principals/teachers of intervention school and/or staffs of The Boys' and Girls' Clubs Association in partnership with HKU research team who organize plan or implement the project
  2. Adults aged 18 or above
  3. Chinese speaking
  4. Intact verbal and hearing abilities for interpersonal communication
  5. Reading and writing abilities for questionnaire/individual in-depth interviews completion

Exclusion Criteria:

* Students who cannot read Chinese

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in the concept of Sharing, Mind and Enjoyment (SME) for adolescents and their family members. | T1: before the 1st Joyful Adventure Day (baseline); T3: after the 2nd Joyful Adventure Day (1-month after baseline); T4: 3-month after baseline
  The outcome-based questionnaire will be used to evaluate participants' frequency of performing the suggested Sharing, Mind and Enjoyment (SME) related behaviors from baseline to three-month after baseline.

SECONDARY OUTCOMES:
Changes in the knowledge and understanding about mental health for adolescents and their family members. | T1: before the 1st Joyful Adventure Day (baseline); T2: immediately after the 1st Joyful Adventure Day ( post intervention ); T3: after the 2nd Joyful Adventure Day (1-month after baseline); T4: 4-month after baseline
  The outcome-based questionnaire will be used to evaluate participants' knowledge and understanding about anxiety disorder from baseline to three-month after baseline.
Changes in personal happiness from baseline to three-month after baseline | T1: before the 1st Joyful Adventure Day (baseline); T3: after the 2nd Joyful Adventure Day (1-month after baseline); T4: 3-month after baseline
  Personal happiness will be assessed by Subjective Happiness Scale (SHS). SHS was rated on 7-point scale with 1 indicating not happiness at all and 7 indicating extreme happiness. To score the scale, the 4th item will be coded reversely and mean of the 4 items will be computed.
Changes in mental well-being from baseline to three-month after baseline. | T1: before the 1st Joyful Adventure Day (baseline); T3: after the 2nd Joyful Adventure Day (1-month after baseline); T4: 3-month after baseline
  Mental well-being will be assessed by validated Chinese version of 7-item Warwick Edinburgh Well-being Scale. Each item ranges from 1 to 5 and the scale will be scored by first summing the score for each of the 7 items and then transforming the total score for each person according to a conversion table.
Changes in individual and family health from baseline to three-month after baseline | T1: before the 1st Joyful Adventure Day (baseline); T3: after the 2nd Joyful Adventure Day (1-month after baseline); T4: 3-month after baseline
  Self-perceived health, happiness and harmony at the individual and family level will be assessed by a 0-10 score at 3 time points
Satisfaction toward Joyful Adventure Day Project | T2: immediately after the 1st Joyful Adventure Day ( post intervention ); T3: after the 2nd Joyful Adventure Day (1-month after baseline); T4: 3-month after baseline
  Satisfaction towards the adventure games, short interactive talk on SME and physical activity diary will be assessed by programme evaluation measure
The social impact of the community-based engagement project | T4: 3-month after baseline
  The social impact of the community-based engagement project will be The satisfaction, ratings and opinions on Joyful Adventure Day programme of school principal/teacher/community partner in the intervention group will be assessed qualitatively (individual in-depth interviews)
The process of community based intervention programme | up to 3 months
  The process evaluation on-site observation questionnaire will be used to assess the process of the community-based intervention programs.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel, Sai Yin Ho, Dr., Principal Investigator — Associate Professor
Locations (1):
- School of Public Health, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No